CLINICAL TRIAL: NCT01909531
Title: Deep Brain Stimulation (DBS) Data Base Study
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Responsible Party: Sponsor
Other Study IDs: 12BN136
Record Dates: First submitted 2013-07-24; First posted 2013-07-26 (Estimated); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Parkinson's Disease; Essential Tremor
Keywords: Deep Brain Stimulation; Parkinsons Disease; Essential Tremor; Asleep DBS
MeSH Terms: conditions — Parkinson Disease; Essential Tremor

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary goal of this study is to evaluate and compare outcomes, trends, and effectiveness of both awake and asleep Deep Brain Stimulation (DBS) surgical treatments, target selection, targeting accuracy and outcomes in patients with Parkinson's disease and Essential tremor.

DETAILED DESCRIPTION:
Deep Brain Stimulation (DBS) surgery is a treatment that can improve some of the motor symptoms associated with several movement disorder diseases. DBS is recommended for patients with Parkinson's disease who respond well to medication, but still experience frequent wearing off of medications with return of symptoms. Patients may also be experiencing troubling medication side effects such as dyskinesias, sleepiness, hallucinations, confusion, and behavioral/personality changes. DBS is also used for patients with Essential tremor who have undergone long trials of medication therapy and are still symptomatic. The goal of DBS surgery is to capture that best response to medication and hold it through the day. The Food and Drug Administration (FDA) approved DBS as a treatment for essential tremor in 1997 and for Parkinson's disease in 2002.

The goal of DBS surgery is to improve the quality of life of patients and their families by reducing motor symptoms such as slowness, stiffness and tremor and possibly reducing medication. In order to help with our understanding of its effects, we will collect information on patients who will be undergoing or have undergone DBS surgery.

St. Joseph's Hospital and Medical Center / Barrow Neurological Institute is one of only a few hospitals in the United States offering a new procedure known as asleep DBS surgery, performed under general anesthesia, as well as the traditional awake DBS procedure; therefore it is important that this new asleep surgery option be studied and compared to awake DBS surgery.

Objectives include:

* Comparison of data collected for both the awake and asleep DBS procedures during the pre-operative and post-operative periods including testing, diagnosis, surgical treatment, target accuracy, complications, motor function and quality of life outcomes.
* Comparison of the differential effects of STN and GPi DBS on gait and balance control
* Investigate the effects of DBS on the saccadic eye movements.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis for Parkinson's Disease or Essential Tremor
* Subject has undergone DBS surgery

Exclusion Criteria:

* Clinical diagnosis for Parkinson's Disease or Essential Tremor
* Subject has not undergone DBS surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's Disease or Essential Tremor who have undergone either awake or asleep DBS surgery performed by Francisco A. Ponce, MD
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2013-04; Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Data Comparison | Pre-operative through 6 months post operative
  Data comparison for pre-operative testing, diagnosis, surgical treatment, target accuracy, complications and outcomes for patients undergoing DBS surgery will be analyzed.

SECONDARY OUTCOMES:
Quantitative Evaluation of Balance and Gait | Pre-operative through 6 months post-operative
  For the quantitative evaluation of gait and balance control, different parameters of gait and balance will be obtained non-invasively during pre- and post-surgical clinical evaluation sessions. For this data collection, patients will be asked to perform many trials of quiet standing (eyes open and eyes closed conditions), postural shifts, stepping-in-place, and regular and tandem walking. These data will be obtained using a portable gait system (consisted of small light-weight sensors) and force plate setup. During balance tests, the patients will be asked to hold on to railings in case of loss of balance and asked to wear gait belt during these evaluations. A member of the research team will be close to the patient to hold them in case of any loss of balance to avoid falls.

OTHER OUTCOMES:
Quantitative Evaluation of Saccadic Eye Movements | Pre-operartive - 6 months post-operative
  Non-invasively record eye movements when patients follow target (light dot on a light bar placed in front of the patients) that jumps, moves back and forth, fixation on target, etc. This data collection will be obtained in a seated position.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco A Ponce, MD, Principal Investigator — St. Joseph's Hospital & Medical Center / Barrow Neurological Institute
Locations (1):
- St. Joseph's Hospital & Medical Center / Barrow Neurological Institute, Phoenix, Arizona, United States